CLINICAL TRIAL: NCT00858039
Title: Prediction of Cardiotoxicity Using Serum N-terminal Pro-B-type Natriuretic Peptide in Breast Cancer Patients Receiving Adjuvant Trastuzumab
Brief Title: Cardiotoxicity of Adjuvant Trastuzumab
Acronym: CATS
Status: Completed | Type: Observational
Sponsor: Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Principal Investigator, Shom Goel, Breast Oncology Fellow, Royal Prince Alfred Hospital, Sydney, Australia
Other Study IDs: X08-0296
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Breast Neoplasms; Heart Failure
MeSH Terms: conditions — Breast Neoplasms; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human serum Human whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Her-2 positive ESBC

SUMMARY:
Trastuzumab (Herceptin®) increases the chances of cure in patients with Her-2 overexpressing early breast cancer. Unfortunately, both the chemotherapy drugs used in this setting (anthracyclines) and trastuzumab are known to cause cardiac dysfunction in a proportion of patients. Patients who develop heart problems when taking trastuzumab might have to stop this treatment, which could jeopardise their chances of cure. N-terminal pro-B-type natriuretic peptide (NT pro-BNP) is a cardiac biomarker that is measured in the blood, the levels of which have been shown to indicate the presence of heart failure. Some early research has suggested that there may be a correlation between elevated NT pro-BNP and heart damage due to cancer chemotherapy and also trastuzumab. Troponin is another substance measured in the blood that can indicate heart damage. Finally, certain variations in an individual's genetic makeup (called polymorphisms) could put them at increased risk of heart damage from trastuzumab. Here we are studying whether any of these factors (NT pro-BNP levels, troponin levels, or certain genetic polymorphisms) can accurately predict who is at highest risk of trastuzumab-related cardiotoxicity.

The principal aim of this study is to evaluate the utility of NT pro-BNP as a predictive biomarker for the development of trastuzumab related cardiotoxicity (TRC). The investigators will also examine if single nucleotide polymorphisms in the HER2 gene or Fc-gamma-receptor genes predict for TRC.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years or older
* Histologically confirmed, completely excised invasive breast cancer with Her-2 overexpression
* Primary surgery less than twelve weeks prior to registration
* LVEF>50% as assessed by transthoracic echocardiogram or gated heart pool scan
* Eastern Cooperative Oncology Group Performance Status 0-2
* Adjuvant systemic treatment plan comprises at least three cycles of anthracycline chemotherapy AND 52 weeks of trastuzumab
* Before patient registration, informed consent must be given according to local regulations.

Exclusion Criteria:

* Pregnancy
* Distant metastases from breast cancer
* Any systemic chemotherapy prior to study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to tertiary referral medical oncology clinics
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2009-02; Primary Completion 2013-07 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cardiotoxicity (Cardiac death; grade 3/4 arrhythmia or ischaemia; NYHA Class 3 or 4 heart failure decline in LVEF by >10% to a level <55%; decline in LVEF by >5% to a level <50%) | Until 6 months after completing trastuzumab

CONTACTS AND LOCATIONS:
Overall Officials: Jane Beith, MBBS FRACP PhD, Study Director — Sydney South West Area Health Service (Royal Prince Alfred Hospital)
Locations (15):
- Australia (15):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal North Shore Private Hospital, Sydney, New South Wales
  - Sydney Haematology Oncology Clinic, Sydney, New South Wales
  - Concord Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Bankstown Hospital, Sydney, New South Wales
  - St George Private Hospital, Sydney, New South Wales
  - Sutherland Hospital, Sydney, New South Wales
  - Macarthur Cancer Therapy Centre, Sydney, New South Wales
  - Nepean Cancer Care Centre, Sydney, New South Wales
  - Tweed Hospital, Tweed Heads, New South Wales
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Andrew Love Cancer Centre, Geelong, Victoria
  - Warnambool Hospital, Warrnambool, Victoria
  - The Mount Hospital, Perth, Western Australia

REFERENCES:
- [Derived] Goel S, Liu J, Guo H, Barry W, Bell R, Murray B, Lynch J, Bastick P, Chantrill L, Kiely BE, Abdi E, Rutovitz J, Asghari R, Sullivan A, Harrison M, Kohonen-Corish M, Beith J. Decline in Left Ventricular Ejection Fraction Following Anthracyclines Predicts Trastuzumab Cardiotoxicity. JACC Heart Fail. 2019 Sep;7(9):795-804. doi: 10.1016/j.jchf.2019.04.014. Epub 2019 Aug 7. PMID 31401102